CLINICAL TRIAL: NCT00644319
Title: A 2 x 2 Factorial Trial to Assess Whether Non-Steroidal Anti-Inflammatory Analgesics and Small Bore Chest Tubes Are Less Painful Than Opiate Analgesics and a Large Bore Chest Tubes in Pleurodesis for Malignant Pleural Effusion [TIME1]
Brief Title: Ibuprofen or Morphine in Treating Pain in Patients Undergoing Pleurodesis for Malignant Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford University Hospitals NHS Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000590072; RADCLIFFE-TIME1; ISRCTN33288337; EUDRACT 2006-005226-31; EU-20829; UKCRN 4035
Record Dates: First submitted 2008-03-25; First posted 2008-03-26 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Metastatic Cancer
Keywords: malignant pleural effusion
MeSH Terms: conditions — Neoplasm Metastasis; Pleural Effusion, Malignant | interventions — Ibuprofen; Morphine; Pleurodesis

INTERVENTIONS:
Drug: ibuprofen
Drug: morphine sulfate
Procedure: management of therapy complications
Procedure: pleurodesis

SUMMARY:
RATIONALE: Morphine and ibuprofen help lessen pain caused by pleurodesis. It is not yet known whether one drug is more effective than the other in lessening pleurodesis-related pain or whether the size of the chest drain tube affects pain.

PURPOSE: This randomized clinical trial is studying ibuprofen to see how well it works compared with morphine in treating pain in patients undergoing pleurodesis for malignant pleural effusion.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of a non-steroidal based regimen comprising ibuprofen in decreasing post-pleurodesis pain as compared to an opiate-based regimen comprising morphine sulfate in patients with malignant pleural effusion.
* To evaluate whether chest drain size influences the amount of post-pleurodesis pain.

OUTLINE: This is a multicenter study. Patients are stratified according to histological tissue type (mesothelioma vs non-mesothelioma) and thoracoscopic procedure. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients undergo pleurodesis after placement of a large bore chest drain (24F) on day 0 and receive oral ibuprofen 3 times daily for 3 days. The chest tube is removed on day 3.
* Arm II: Patients undergo pleurodesis after placement of a small bore chest drain (12F) on day 0 and receive oral ibuprofen 3 times daily for 3 days. The chest tube is removed on day 3.
* Arm III: Patients undergo pleurodesis after placement of a large bore chest drain (24F) on day 0 and receive oral morphine sulfate 4 times daily for 3 days. The chest tube is removed on day 3.
* Arm IV: Patients undergo pleurodesis after placement of a small bore chest drain (12F) on day 0 and receive oral morphine sulfate 4 times daily for 3 days. The chest tube is removed on day 3.

All patients will receive regular background analgesia comprising paracetamol 4 times daily on days 0-3. Patients not adequately treated with these regimens may also receive rescue analgesia comprising morphine sulfate IV on days 0-3.

After completion of study treatment, patients are followed at 1, 3, and 6 months, and periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignant pleural effusion requiring pleurodesis confirmed by 1 of the following:

  * Histologically proven pleural malignancy
  * Typical features of pleural malignancy seen on direct vision during thoracoscopy
  * Pleural effusion in the context of histologically proven cancer elsewhere
* No primary lymphoma or small cell lung carcinoma
* All patients undergoing thoracoscopy for suspected malignant pleural effusion are eligible

PATIENT CHARACTERISTICS:

* Life expectancy > 1 month
* Not pregnant or nursing
* No history of GI bleeding or untreated peptic ulceration
* No known sensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), opiates, or paracetamol
* No hypercapnic respiratory failure
* No known intravenous drug abuse
* No severe renal or liver disease
* No known bleeding diathesis
* Able to give informed consent

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior and no concurrent corticosteroid therapy
* No concurrent warfarin therapy
* No other concurrent analgesics

  * Analgesics used as a breakthrough regimen are allowed from trial entry to tube withdrawal at day 3 post-pleurodesis (i.e., regular paracetamol, assigned study analgesia, and breakthrough medication only, including opiate slow release patches)
* No concurrent enrollment on another clinical study

  * Patients may participate in other trials immediately after completion of current trial, excluding those involving further pleural procedures or analgesia trials in which patients must wait at least 3 months after completion of current trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Average pain score over 72 hours post pleurodesis (total pain relief score) by a Visual Analogue Scale of pain relief and pain intensity every 6 hours
Pleurodesis success at 3 months post randomization (time to relapse of pleural effusion, censored for survival)

SECONDARY OUTCOMES:
Presence of chronic chest pain on the side of the pleurodesis at 6 weeks and 3 months post randomization
Change in hemoglobin and white cell count from day 0 to day 3
Change in renal function and liver function (i.e., ALT or AST, bilirubin, albumin, and alk phos) from day 0 to day 3
Change in Inflammatory markers from day 0 and day 3 (e.g., CRP, WCC) from day 0 to day 3
Change in alveolar PO2-arterial PO2 (A-a) gradient (on air) on day 0 and day 3
Continuous oximetry monitoring from day 0 to day 3 (on air unless saturation < 90%)
Average conscious level measured by Glasgow Coma scale from day 0 to day 3
Drug- and talc-related adverse reactions
Complications from chest drain insertion
Presence of chronic chest wall pain assessed at all follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Robert Davies, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Radcliffe Hospital, Oxford, England, United Kingdom